CLINICAL TRIAL: NCT05164263
Title: Real World Safety & Efficacy Experience of Empagliflozin With or Without Metformin in Patients With Type II Diabetes Mellitus
Brief Title: Real World Safety & Efficacy Experience of Empagliflozin With or Without Metformin in T2DM Patients - EASE Study
Acronym: EASE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTZ-DM-003-21
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type II Diabetes Mellitus; Efficacy, Self; Safety Issues
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, observational, single arm, multi-center, post-marketing surveillance study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin naive uncontrolled T2DM on oral anti-diabetics & lifestyle modifications for 3 months (Experimental): Type 2 diabetic males & females between 18-65 years.
  * HbA1c: 7.0% - 10%
  * eGFR ˃60 mL/min/1.73m2.
  * Patient who will give informed consent
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin + Metformin (Diampa™-M): 5mg+500mg, 5mg+850mg, 5mg+1000mg, 12.5mg+1000mg, 12.5mg+500mg, 12.5mg+ 850mg Empagliflozin Alone (Diampa™): 10mg, 25mg

SUMMARY:
Study Objective To evaluate the safety and tolerability of Empagliflozin with or without metformin in patients with Type II Diabetes Mellitus in the Pakistani population.

Study design Open-label, prospective, observational, single arm, multi-center, post-marketing surveillance study.

Sample size The estimated sample size will be n=156. Duration of study 12 months (data lock point will be completion of 6 months' follow-up from the time of last patient's enrollment date) Safety Assessment: Patient will be monitored for Hypoglycemia, Dehydration, Hypotension, Urinary Tract Infections, Fungal Infections, Nausea, Vomiting, Diarrhea, Abdominal Discomfort, Flatulence, Asthenia, Indigestion and Other side effects (if any).

Follow up visits: After recruitment, patient is supposed to have three visits for follow-ups.

Visit 1: 4 to 6 weeks of initiation of therapy. Visit 02: At 12 weeks of initiation of therapy. Visit 03: At 24 weeks of initiation of therapy.

LABORATORY TESTING:

Reputable Lab is considered for laboratory testing of diabetes patients i.e. HbA1C%, FBG, RFT and urine R/E. The certified clinical lab will be responsible for receiving and analyzing clinical sample. Patients will have special discount of upto 50% for study related laboratory investigations.

Where in Urine Routine Examination (Urine R/E), we consider as follows:

* Visual Examination:

  * Urine color: Normal (Yellow), Pale Yellow, Dark Yellow, Brown, Red or Pink or any other.
  * Urine clarity: Clear, slightly Cloudy, cloudy or turbidity
* Chemical Examination:

  * Specific gravity
  * pH
  * Bilirubin
  * Urobilinogen
  * Protein
  * Ketone
  * Leukocyte Esterase
* Microscopic Examination:

  * Red Blood Cells:
  * Epithelial Cells:
  * Amorphous:
  * Pus Cells
  * Bacteria
  * Yeast
  * Casts
  * Crystals

Where in Renal Function Test (RFT), we consider as follows:

* Blood Urea Nitrogen (BUN): mg/dL
* Serum Creatinine: mg/dL
* Estimated Glomerular Filtration Rate (eGFR): mL/min/1.73 m2

ELIGIBILITY:
Inclusion Criteria:

Patient with T2DM between 18 to 65 years with HbA1C 7% - 10%, who can give informed consent. Patient uncontrolled on oral antidiabetics and lifestyle modification for at least 3 months. Patient who are empagliflozin naive. eGFR ˃60 mL/min/1.73m2.

Exclusion Criteria:

Type 1 diabetes, History of recurrent urinary tract infection (UTI), fungal infection, renal and/or hepatic dysfunctions, where RFT and Urine R/E is abnormal, Diabetic Ketoacidosis and/or hyperosmolar hyperglycemic state, severe hypoglycemia, Pregnant or lactating women, Pancreatitis, any serious complications or hypersensitivity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
SAFETY and TOLERABILITY Outcomes | 6 months
  Frequency of adverse events, serious adverse events during the course of study follow-up. Percentage of patients who tolerate empagliflozin.

SECONDARY OUTCOMES:
Efficacy outcomes | 6 months
  Change from baseline in HbA1c% and fasting plasma glucose to the last-observation on treatment. Change from baseline in bodyweight & other study parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Umar Wahab, Principal Investigator — Umar Diabetes Foundation
Locations (6):
- Kabul University of Medical Sciences(KUMS), Kabul, Afghanistan, Afghanistan
- Agha Khan univeristy hospital, Nairobi, Kenya, Kenya
- Lagos University Teaching Hospital, Lagos, Nigeria, Nigeria
- Umar Diabetes Foundation, Islamabad, Pakistan
- Sri Lanka (2):
  - National hospital Sri Lanka, Colombo, Colombo
  - NHK, Kandy, Kandy

IPD SHARING:
Plan to Share IPD: No
Upon request

REFERENCES:
- [Background] Ferrannini E, Mark M, Mayoux E. CV Protection in the EMPA-REG OUTCOME Trial: A "Thrifty Substrate" Hypothesis. Diabetes Care. 2016 Jul;39(7):1108-14. doi: 10.2337/dc16-0330. PMID 27289126
- [Background] Barnett AH, Mithal A, Manassie J, Jones R, Rattunde H, Woerle HJ, Broedl UC; EMPA-REG RENAL trial investigators. Efficacy and safety of empagliflozin added to existing antidiabetes treatment in patients with type 2 diabetes and chronic kidney disease: a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2014 May;2(5):369-84. doi: 10.1016/S2213-8587(13)70208-0. Epub 2014 Jan 24. PMID 24795251